CLINICAL TRIAL: NCT05299099
Title: A Randomized, Open-label, Multi-center Phase III Clinical Trial to Evaluate the Safety and Efficacy of IN-C006 Inj. Compared With RCN301 in Postoperative Patients Requiring Central Parenteral Nutrition
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of IN-C006 Inj. Compared With RCN301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IN_CPN_301
Record Dates: First submitted 2022-03-02; First posted 2022-03-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-02

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-C006 inj. (Experimental): IN-C006 inj. 1970 mL
  Interventions: Drug: IN-C006 inj.
- RCN301 (Active Comparator): RCN301 1820 mL
  Interventions: Drug: RCN301

INTERVENTIONS:
Drug: IN-C006 inj. — IN-C006 will be injected continuously for 3 days.
  Other Names: IN-C006 inj
  Arms: IN-C006 inj.
Drug: RCN301 — RCN301 will be injected continuously for 3 days.
  Arms: RCN301

SUMMARY:
This study is designed to evaluate the safety and efficacy of IN-C006 inj. and RCN301 in postoperative patients requiring central parenteral nutrition.

DETAILED DESCRIPTION:
This study is a randomized, open-label, phase 3 design. The subject will be assigned to one of the two treatment groups (IN-C006 inj. or RCN301)

ELIGIBILITY:
Inclusion Criteria:

* Age over 19 at the time of obtaining the informed consent form
* Requiring over 3 days of parenteral nutrition via a central vein after an operation
* BMI 16 ~ 30 kg/㎡

Exclusion Criteria:

* Has received parenteral nutrition within 7 days of screening
* Severe dyslipidemia
* Uncontrolled diabetes
* Clinically significant liver disease
* Clinically significant kidney disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse drug reaction rate | Day 1 to Day 4
  Rate of treatment-related adverse events as assessed by CTCAE v5.0 and investigator's evaluation

SECONDARY OUTCOMES:
Change in nutritional management parameters | Day 1 to Day 4
  Nitrogen balance(Nitrogen intake-Nitrogen out), Prealbumin(mg/L), Albumin(g/dL), Transferrin(mg/dL)
Change in inflammation parameters | Day 1 to Day 4
  hs-CRP(mg/L), TNF-α(pg/mL), IL-6(pg/mL)
Change in fatty acid profile | Day 1 to Day 4
  LA(ug/mL), AA(ug/mL), EPA(ug/mL), DHA(ug/mL)
Incidence of Adverse event | Day 1 to Day 4
  Rate of adverse events as assessed by CTCAE v5.0 and investigator's evaluation
Change in laboratory parameters | Day 1 to Day 4
  Hematology, Blood chemistry, Blood coagulation test, Urinalysis
Change in vital sign | Day 1 to Day 4
  Blood pressure(mmHg), pulse rate(rate), body temperature(℃) and respiratory rate(rate)
Normal and abnormal change in physical examination | Day 1 to Day 4
  General Appearance, HEENT (Head, Eyes, Ears, Nose, Throat), Skin (including hair, nails), Respiratory, Cardiovascular, Chest/Lungs/Breast, Abdominal/Gastrointestinal, Musculoskeletal, Extremities/Joint, Neurological/Psychological, Lymph nodes, Rectal/Pelvic/Genitalia, Other

CONTACTS AND LOCATIONS:
Overall Officials: Do Joong PARK, Study Chair — Seoul National Univerity Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No